CLINICAL TRIAL: NCT03195634
Title: WFA+M2BP in Evaluation of Portal Hypertension and Clinical Outcome in Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Shanghai Changzheng Hospital
Other Study IDs: CZXH0021
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HVPG group: When HVPG > 12 mmHg, patients would be treated with carvedilol at an initial dose of 6.25 mg once-daily that was adjusted over 5-7 days to the maximum tolerated dose, keeping heart rate >55 beats per minute, or up to 12.5 mg/day.
  After about 8 weeks, the patients treated with carvedilol will received the second HVPG monitoring wether achieved a decrease in HVPG below 12 mm Hg or>20% from baseline.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — an initial dose of 6.25 mg once-daily that was adjusted over 5-7 days to the maximum tolerated dose, keeping heart rate >55 beats per minute, or up to 12.5 mg/day

SUMMARY:
Portal hypertension is a common complication of chronic liver diseases and is responsible for most clinical consequences of cirrhosis. measurement of the hepatic venous pressure gradient(HVPG) is the gold standard for evaluating the presence and severity of portal hypertension, this technique is considered invasive and is not routinely performed in all centers. Wisteria floribunda agglutinin-positive human Mac-2 binding protein (WFA+-M2BP) is a secreted N-glycoprotein, which has been reported as a novel marker in assessing liver fibrosis.However, the correlation of WFA+-M2BP with HVPG is unclear.The aim of this study was to explore the relationship between WFA+-M2BP and HVPG.

DETAILED DESCRIPTION:
Portal hypertension is a common complication of chronic liver diseases and is responsible for most clinical consequences of cirrhosis. Accurate assessment of portal hypertension is essential for strategy of treatment and judgement of prognosis. Although measurement of the hepatic venous pressure gradient(HVPG) is the gold standard for evaluating the presence and severity of portal hypertension, this technique is considered invasive and is not routinely performed in all centers. Therefore, it is urgent to explore a noninvasive assessment of portal hypertension.

Wisteria floribunda agglutinin-positive human Mac-2 binding protein (WFA+-M2BP) is a secreted N-glycoprotein, which has been reported as a novel marker in assessing liver fibrosis. Recently, a retrospective study investigated the role of WFA+-M2BP in assessing the degree of liver cirrhosis and predicting mortality. However, the correlation of WFA+-M2BP with HVPG is unclear. And the role of WFA+-M2BP in predicting the clinical outcome of liver fibrosis patients is needed to be further evaluated.

The aim of this study was to explore the relationship between WFA+-M2BP and HVPG, as well as its predictive ability of complication rate, including large varices, bleed status, and ascites, and liver disease-related mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients agreed to sign the informed consents
2. Patients aged 18-80 years,males or females
3. Patients with liver cirrhosis was diagnosed by previous liver biopsy or by compatible clinical, biochemical, and ultrasonographic/CT/MRI findings.
4. Patients were not treated with nonselective β-blockers(propranolol or carvedilol ) within previous 3 months

Exclusion Criteria:

1. Uncontrolled hypertension, diabetes or other serious cardiac problems（NYHA class IV）and pulmonary disease
2. Severe renal function injury(serum creatinine≥1.2 fold of upper limits of normal)
3. Conformed or highly suspicious diagnosis of liver malignant tumors or concomitant disease with reduced life expectancy
4. Acute hepatic failure or acute on chronic liver failure(ACLF)
5. Human immunodeficiency virus(HIV) infection
6. Previous portosystemic shunt
7. After liver transplantation
8. Pregnancy and breastfeeding
9. With contraindications of intervention surgery(hypersensitivity to iodinated contrast media, puncture site infection, severe coagulation defects, uncontrolled hyperthyroidism and multiple myeloma)
10. Participated in other drug clinical trails within 3 months
11. The researchers thought it was not suitable for this clinical trail

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 2017 to March 2018, patients with cirrhosis admitted to either of the two participating hospitals were consecutively enrolled.
  Hospitals: Shanghai Changzheng hospital and Shandong Provincial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of portal pressure (PP) | 3 months
  portal pressure (PP) will be estimated from the hepatic venous pressure gradient(HVPG)
serum WFA+-M2BP levels | 3 months
  serum WFA+-M2BP levels

SECONDARY OUTCOMES:
number of death or liver transplantation | up to 1 year
  number of death or liver transplantation
complications of cirrhosis | up to 1 year
  large varices, bleed status and ascites

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, MD, Principal Investigator — Department of Gastroenterology, Changzheng Hospital, Second Military Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: No